CLINICAL TRIAL: NCT04464226
Title: An Open-label, Single Arm, Roll-over Study to Provide Continued Treatment With Darolutamide in Participants Who Were Enrolled in Previous Bayer Sponsored Studies
Brief Title: Study to Continue Treatment With Darolutamide in Patients Who Have Been Participating in Previous Darolutamide Studies Supported by Bayer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20321; 2019-003618-15 (EudraCT Number)
Record Dates: First submitted 2020-07-07; First posted 2020-07-09 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Cancer
Keywords: Roll-Over Study
MeSH Terms: conditions — Neoplasms | interventions — darolutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Darolutamide (BAY1841788) (Experimental): Participants enrolled in the current study will use the dose they were assigned to in the feeder study they come from.
  Interventions: Drug: Darolutamide (Nubeqa, BAY1841788)

INTERVENTIONS:
Drug: Darolutamide (Nubeqa, BAY1841788) — Participants will continue receiving darolutamide treatment at the dose level and schedule of administration previously assigned in the feeder study.
  Other Names: ODM-201

SUMMARY:
The aim of this study is to provide darolutamide treatment to patients who participated in a previous study with darolutamide supported by Bayer and the treating doctor considers that the continuation of the treatment with darolutamide to be beneficial. Patients will be carried over from the previous studies and continue in this study with darolutamide treatment on the same dosage. They will also return to the study centers for doctor's visits as often as they did in the previous study.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
* Participants enrolled in any Bayer-sponsored darolutamide feeder study at the time of study closure or primary completion, who are currently receiving darolutamide and are experiencing clinical benefit from treatment.
* Participants who have not met any treatment discontinuation criteria in the feeder study protocol.
* Willingness to continue practicing acceptable methods of birth control during the study.

Exclusion Criteria:

* Participant is unable to comply with the requirements of the study.
* Negative benefit/ risk ratio as determined by the investigator.
* Meet any criteria for treatment discontinuation of the feeder study the participant is coming from.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 402 (Estimated)
Dates: Start 2020-10-20 (Actual); Primary Completion 2028-06-26 (Estimated); Study Completion 2028-06-26 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) | Up to 4 years
Incidence of treatment-emergent serious adverse events (TESAEs) | Up to 4 years
Incidence of drug-related TEAEs | Up to 4 years
Incidence of drug-related TESAEs | Up to 4 years

SECONDARY OUTCOMES:
Number of dose modifications | Up to 4 years

CONTACTS AND LOCATIONS:
Locations (380):
- United States (45):
  - Urology Centers of Alabama, PC, Homewood, Alabama
  - Ironwood Cancer and Research Centers - Chandler I, Chandler, Arizona
  - City of Hope National Medical Center, Duarte, California
  - Tower Urology, Los Angeles, California
  - VA Greater Los Angeles Healthcare System, Los Angeles, California
  - Stanford Cancer Center Palo Alto, Palo Alto, California
  - San Diego Clinical Trials, San Diego, California
  - TOI Clinical Research, Whittier, California
  - VA Eastern Colorado Health Care System, Aurora, Colorado
  - The Urology Center Of Colorado, Denver, Colorado
  - Boca Raton Regional Hospital - Oncology, Boca Raton, Florida
  - Advent Health Medical Group Urology, Orlando, Florida
  - Jesse Brown VA Medical Center - Cardiology, Chicago, Illinois
  - Illinois CancerCare - Peoria, Peoria, Illinois
  - First Urology PSC, Jeffersonville, Indiana
  - Norton Cancer Institute - Downtown, Louisville, Kentucky
  - Anne Arundel Health System, Annapolis, Maryland
  - Chesapeake Urology Associates - Towson, Baltimore, Maryland
  - Johns Hopkins Hospital - Pulmonology, Baltimore, Maryland
  - TidalHealth Peninsula Regional, Inc. - Oncology, Salisbury, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Henry Ford Hospital - OB/GYN, Detroit, Michigan
  - St. Vincent Regional Hospital - Oncology, Billings, Montana
  - Urology Cancer Center, PC, Omaha, Nebraska
  - XCancer Omaha, Omaha, Nebraska
  - New Jersey Urology - Voorhees, Voorhees Township, New Jersey
  - New Mexico Cancer Center - Albuquerque, Albuquerque, New Mexico
  - URMC Wilmot Cancer Center, Rochester, New York
  - Associated Medical Professionals of NY, PLLC, Syracuse, New York
  - New York Cancer & Blood Specialists - Eastchester, The Bronx, New York
  - Montefiore Einstein Center for Cancer Care, The Bronx, New York
  - Gabrail Cancer Center, Canton, Ohio
  - The Urology Group - Norwood Surgery Center, Cincinnati, Ohio
  - The Ohio State University - Arthur G James Cancer Hospital and Richard J Solove Research Institute, Columbus, Ohio
  - MidLantic Urology - Bala Cynwyd, Bala-Cynwyd, Pennsylvania
  - Andrews & Patel Associates, Camp Hill, Pennsylvania
  - Charleston Oncology - Downtown, Charleston, South Carolina
  - Bon Secours St. Francis Hospital, Greenville, South Carolina
  - Carolina Urological Research Center, Myrtle Beach, South Carolina
  - Urology Associates, PC, Nashville, Tennessee
  - Urology Clinics of North Texas, Dallas, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Inova Schar Cancer Insitute - Inova Fairfax Hospital, Fairfax, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Providence Regional Cancer Partnership, Everett, Washington
- Centro de Urología, Buenos Aires, Ciudad Auton. de Buenos Aires, Argentina
- Adelaide Cancer Centre Research Pty Ltd, Kurralta Park, South Australia, Australia
- Universitätsklinikum AKH Wien, Vienna, Austria
- Belarus (2):
  - N.N. Alexandrov National Cancer Centre of Belarus - Oncology Department, Lesnoy
  - Minsk City Clinical Oncological Dispensary - Oncology Department, Minsk
- Belgium (6):
  - GZA Ziekenhuizen, Wilrijk, Antwerpen
  - CU Saint-Luc/UZ St-Luc, Bruxelles - Brussel
  - UZ Gent, Ghent
  - AZ Groeninge Campus Kennedylaan, Kortrijk
  - CHU de Liège, Liège
  - CHU UCL Namur, Namur
- Brazil (19):
  - Instituto do Cancer do Ceará, Fortaleza, Ceará
  - Hospital Evangélico de Cachoeiro de Itapemirim, Cachoeiro de Itapemirim, Espírito Santo
  - Hospital São Rafael, Salvador, Estado de Bahia
  - Santa Casa de Misericórdia da Bahia, Salvador, Estado de Bahia
  - Hosp. Araujo Jorge da Associação de Combate ao Câncer, Goiânia, Goiás
  - COT Centro Oncologico do Triangulo Ltda, Uberlândia, Minas Gerais
  - Liga Paranaense de Combate ao Cancer-Hosp Erasto Gaertner, Curitiba, Paraná
  - Liga Norte Riograndense Contra o Cancer | Centro de Pesquisa Clínica, Natal, Rio Grande do Norte
  - Associação Hospitalar Beneficente São Vicente de Paulo, Passo Fundo, Rio Grande do Sul
  - Irmandade Santa Casa de Misericordia de Porto Alegre | Oncology, Porto Alegre, Rio Grande do Sul
  - União Bras. de Edu. e Assist. Hospital São Lucas da PUCRS, Porto Alegre, Rio Grande do Sul
  - Clínica de Neoplasias Litoral Ltda, Itajaí, Santa Catarina
  - Fundacao Pio XII - Hospital de Cancer de Barretos, Barretos/SP, São Paulo
  - Hospital Amaral Carvalho, Jaú, São Paulo
  - Hosp Clínicas Facult. Med. de Ribeirão Preto / USP, Ribeirão Preto, São Paulo
  - IEP São Lucas, São Paulo, São Paulo
  - Instituto do Cancer do Estado de Sao Paulo, São Paulo, São Paulo
  - IBCC - Instituto Brasileiro de Controle do Cancer, São Paulo, São Paulo
  - Inst. de Assistência Médica ao Sérvidor Público Estadual, São Paulo, São Paulo
- Bulgaria (2):
  - Medical Center Kalimat, Sofia
  - Complex Oncology Center - Vratsa, Vratsa
- Canada (10):
  - Prostate Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Nova Scotia Health Authority, Halifax, Nova Scotia
  - G. Kenneth Jansz Medicine Professional Corporation, Burlington, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - London Health Sciences Centre, London, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Princess Margaret Hospital-University Health Network, Toronto, Ontario
  - CIUSSS de l'Estrie- Centre Haute-Yamaska, Granby, Quebec
  - Centre Hospitalier de l'Universite de Montreal (CHUM), Montreal, Quebec
- China (44):
  - The Second Hospital of Anhui medical university, Hefei, Anhui
  - Anhui Provincial Hospital, Hefei City, Anhui Province, Anhui
  - Beijing Cancer Hospital - Oncology Department, Beijing, Beijing Municipality
  - Beijing Hospital, Beijing, Beijing Municipality
  - The First Affiliated hospital of Fujian Medical University, Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - 2nd Affiliated Hosp. of Shantou University Medical College, Shantou, Guangdong
  - Tongji Hosp. of Tongji Med Coll, Huazhong Uni of Sci & Tech., Wuhan, Hubei
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Hunan Cancer Hospital - Oncology Department, Changsha, Hunan
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu
  - NJ Drum Tower Hospital, the Affil Hos of NJ Univ Med School, Nanjing, Jiangsu
  - The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Nantong tumor hospital, Nantong, Jiangsu
  - The 2nd Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The First Affiliated Hospital of NanChang University, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - Liaoning Cancer Hospital and Institute, Shengyang, Liaoning
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Qilu Hosp., Shandong Univ., Jinan, Shandong
  - Yantai Yuhuangding Hospital, Yantai, Shandong
  - Shanxi Medical University - First Hospital, Taiyuan, Shanxi
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - University of Electronic Science & Technology of China - Sichuan Cancer Hospital & Institute (Sichuan Provincial Tumor Hospital), Chengdu, Sichuan
  - Sichuan University West China Hospital, Chengdu, Sichuan
  - ZheJiang Provincial People's Hospital, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - Cancer Hospital, Chinese Academy of Medical Sciences, Beijing
  - Peking University Third Hospital, Beijing
  - Sichuan Academy of Medical Sciences & Sichuan Provincial People's Hospital (SAMSPH), Chengdu
  - Chongqing Cancer Hospital, Chongqing
  - Sun Yat-sen University Cancer Center, Guangzhou
  - Ningbo First Hospital, Ningbo
  - The Affiliated Hospital of Qingdao University, Shandong
  - Fudan University Shanghai Cancer Center - Oncology Department, Shanghai
  - Ruijin Hosp. Shanghai Jiaotong Univ.School of Medicine, Shanghai
  - Zhongshan Hospital, Fudan University - Oncology Department, Shanghai
  - Huadong Hospital, Affiliated to Fudan University, Shanghai
  - Shanghai Tenth People's Hospital, Shanghai
  - Shanghai General Hospital, Shanghai
  - Cancer Hospital Chinese Academy of Medical Sciences, Shenzhen Center, Shenzhen
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin
  - The Second Hospital of Tianjin Medical University, Tianjin
  - ZheJiang Provincial People's Hospital, Zhejiang
- Colombia (3):
  - Hospital Pablo Tobón Uribe, Medellín, Antioquia
  - Oncomédica S.A., Montería, Departamento de Córdoba
  - Fundación Oftalmológica de Santander Carlos Ardila Lule, Floridablanca, Santander Department
- Czechia (6):
  - Masarykuv onkologicky ustav, Brno
  - Nemocnice Jablonec nad Nisou, Jablonec nad Nisou
  - Fakultni nemocnice Kralovske Vinohrady, Prague
  - Urocentrum Praha, s.r.o., Prague
  - Všeobecná fakultní nemocnice v Praze, Prague
  - ANDROGEOS, spol. s r.o., Prague
- Sihtasutus Põhja-Eesti Regionaalhaigla - Onkoloogia- ja hematoloogiakliinik, Tallinn, Estonia
- Finland (7):
  - HUS, Meilahden sairaala, Helsinki, Uusimaa
  - Keski-Suomen sairaala Nova, Jyväskylä
  - Mikkelin keskussairaala, Mikkeli
  - Oulun yliopistollinen sairaala, Oulu
  - Seinäjoen keskussairaala, Seinäjoki
  - Tampere University Hospital, Tampereen yliopistollinen sairaala (TAYS), Tampere
  - Turun yliopistollinen keskussairaala, Turku
- France (20):
  - Centre Hospitalier Universitaire - Angers, Angers
  - Institut Bergonie - Unicancer Nouvelle Aquitaine - Service Oncologie medicale, Bordeaux
  - Clinique Lanroze, Brest
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre d'Oncologie et de Radiologie du Parc, Dijon
  - Institut Paoli-Calmettes - Marseille, Marseille
  - ICM - Institut du Cancer de Montpellier - Val d'Aurelle, Montpellier
  - Centre d'Oncologie de Gentilly, Nancy
  - Hopital Hotel Dieu - Nantes, Nantes
  - Hôpital Saint Louis, Paris
  - HCL - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Hôpital de la Milétrie, Poitiers
  - Institut de Cancerologie Jean Godinot - Departement oncologie medicale, Reims
  - CHU Rennes - Hopital Pontchaillou, Rennes
  - Hôpital Charles Nicolle, Rouen
  - Institut de Cancerologie Ouest - Saint-Herblain, Saint-Herblain
  - Hôpital d'Instruction des Armées Begin, Saint-Mandé
  - Centre Médico-Chirurgical Foch, Suresnes
  - CHU Tours - Hopital Bretonneau, Tours
  - Gustave Roussy - Departement Oncologie-Radiotherapie, Villejuif
- Germany (19):
  - Urologische Gemeinschaftspraxis Carl-Andreas-Meilinger, Emmendingen, Baden-Wurttemberg
  - Universitätsklinikum Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - Urologische GemPraxis Dr. R. Rudolph, Kirchheim unter Teck, Baden-Wurttemberg
  - Urologische Gemeinschaftspraxis Muehlacker, Mühlacker, Baden-Wurttemberg
  - Studienpraxis Urologie, Nürtingen, Baden-Wurttemberg
  - Urologische Gemeinschaftspraxis Dr. Simone Maier, Reutlingen, Baden-Wurttemberg
  - Uniklinik Tübingen / Urologie, Tübingen, Baden-Wurttemberg
  - Universitätsklinikum Ulm, Ulm, Baden-Wurttemberg
  - Universitätsklinikum Erlangen, Erlangen, Bavaria
  - Universitätsklinikum der Johann Wolfgang Goethe Universität, Frankfurt am Main, Hesse
  - Städtisches Klinikum Braunschweig gGmbH, Braunschweig, Lower Saxony
  - Gesundheitszentrum Holzminden, Holzminden, Lower Saxony
  - Heinrich-Heine-Universität Düsseldorf, Düsseldorf, North Rhine-Westphalia
  - Praxis Drs. Tim Schneider /B. Schneider, Mülheim, North Rhine-Westphalia
  - Universitätsklinikum Münster, Münster, North Rhine-Westphalia
  - Uro-Gyn-Zentrum Wall Hr. Dr. Jochen Gleißner, Wuppertal, North Rhine-Westphalia
  - Universitätsmedizin der Johannes Gutenberg Universität Mainz, Mainz, Rhineland-Palatinate
  - Medizinische Fakultät der Otto-von-Guericke Universität, Magdeburg, Saxony-Anhalt
  - Friedrich-Schiller-Uni. Jena, Jena, Thuringia
- Hungary (3):
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Tolna Varmegyei Balassa Janos Korhaz, Szekszárd
  - Zala Varmegyei Szent Rafael Korhaz, Zalaegerszeg
- Israel (3):
  - Clalit Health | Soroka Medical Center - Internal Medicine Department, Beersheba
  - Rabin Medical Center | Beilinson Hospital - Internal Medicine C Department, Petah Tikva
  - Health Corporation of the Ziv Medical Center (R.A.), Safed
- Italy (5):
  - IRCCS Istituto Nazionale Tumori Fondazione Pascale, Napoli, Campania
  - Azienda Ospedaliero Universitaria Parma, Parma, Emilia-Romagna
  - Azienda Ospedaliero-Universitaria San Luigi Gonzaga - Oncologia Medica, Orbassano, Piedmont
  - Istituto Di Candiolo Fondazione Del Piemonte Per L'Oncologia IRCCS, Turin, Piedmont
  - Istituto Oncologico Veneto_Padova - UOC Oncologia 1, Padua, Veneto
- Japan (38):
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - Asahi General Hospital, Asahi, Chiba
  - Toho University Sakura Medical Center, Sakura, Chiba
  - Gunma University Hospital, Maebashi, Gunma
  - Sapporo Medical University Hospital, Sapporo, Hokkaido
  - Kobe University Hospital, Kobe, Hyōgo
  - National hospital Organization Mito Medical Center, Higashiibaraki, Ibaraki
  - Kitasato University Hospital, Sagamihara, Kanagawa
  - Yokohama City University Medical Center, Yokohama, Kanagawa
  - Yokosuka Kyosai Hospital, Yokosuka, Kanagawa
  - Mie University Hospital, Tsu, Mie-ken
  - National Hospital Organization Shinshu Ueda Medical Center, Ueda, Nagano
  - Oita University Hospital, Yufu, Oita Prefecture
  - Osaka International Cancer Institute, Osaka, Osaka
  - Kindai University Hospital, Sayama, Osaka
  - The University of Osaka Hospital, Suita, Osaka
  - Hamamatsu University Hospital, Hamamatsu, Shizuoka
  - Saiseikai Utsunomiya Hospital, Utsunomiya, Tochigi
  - Nippon Medical School Hospital, Bunkyo-Ku, Tokyo
  - Juntendo University Hospital, Bunkyo-ku, Tokyo
  - Tokyo Metropolitan Institute for Geriatrics and Gerontology, Itabashi-ku, Tokyo
  - Kyorin University Hospital, Mitaka, Tokyo
  - Tokyo Metropolitan Police Hospital, Nakano-ku, Tokyo
  - Keio University Hospital, Shinjuku-ku, Tokyo
  - The Fraternity Memorial Hospital, Sumida-ku, Tokyo
  - Tottori University Hospital, Yonago, Tottori
  - Yamaguchi University Hospital, Ube, Yamaguchi
  - Chiba Cancer Center, Chiba
  - Gifu Prefectural General Medical Center, Gifu
  - Hiroshima City Hiroshima Citizens Hospital, Hiroshima
  - National Cancer Center Hospital East, Kashiwa
  - National Hospital Organization Kumamoto Medical Center, Kumamoto
  - University of Miyazaki Hospital, Miyazaki
  - Nagasaki University Hospital, Nagasaki
  - Osaka Metropolitan University Hospital, Osaka
  - Osaka General Medical Center, Osaka
  - Toyama University Hospital, Toyama
  - Wakayama Medical University Hospital, Wakayama
- Latvia (6):
  - Daugavpils Regional Hospital, Daugavpils
  - Litavniece Dzintra practice in urology and oncological chem., Liepāja
  - P. Stradins Clinical University Hospital, Riga
  - AS "Association of Health Centers" polyclinic "Elite", Riga
  - Riga East Clinical University Hospital "Gailezers", Riga
  - Vidzemes Hospital, Valmiera
- Lithuania (4):
  - Hospital of LT University of Health Sciences Kaunas Clinics, Kaunas
  - PI Klaipedos University Hospital, Klaipėda
  - National Cancer Institute, Vilnius
  - Vilnius University Hospital Santaros Klinikos, Vilnius
- Mexico (2):
  - Hospital Universitario "José Eleuterio González", Monterrey, Nuevo León
  - INBIOMEDyC Querétaro, Querétaro City, Querétaro
- Netherlands (8):
  - Nederlands Kanker Instituut, Amsterdam
  - Academisch Medisch Centrum (AMC), Amsterdam
  - Albert Schweitzer Ziekenhuis | Dordwijk - Cardiology Department, Dordrecht
  - Zuyderland Medical Centre | Internal Medicine Department, Geleen
  - Tergooi MC | Hilversum - Wetenschapsbureau, Hilversum
  - Spaarne Gasthuis, Hoofddorp
  - HagaZiekenhuis, The Hague
  - ETZ TweeSteden Ziekenhuis (vh Maria Ziekenhuis), Tilburg
- Peru (3):
  - Centro Médico Monte Carmelo - Oncology Department, La Victoria, Arequipa
  - Hospital Central de la Fuerza Aerea del Perú, Lima
  - Instituto Peruano de Oncología & Radioterapia - Oncologia SA - Oncology Department, Lima
- Poland (10):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - ETG Network Spolka z o.o., Lodz
  - KO-MED Centra Kliniczne Lublin II, Lublin
  - Europejskie Centrum Zdrowia Otwock, Szpital im. F. Chopina, Otwock
  - SPZOZ Wojewodzki Szpital Specjalistyczny nr 3, Rybnik
  - Urologica Praktyka Lekarska Adam Marcheluk, Siedlce
  - Mazowiecki Szpital Onkologiczny, Waliszew
  - Centrum Onkologii - Instytut im. M.Sklodowskiej-Curie, Warsaw
  - Szpital Grochowski im. dr.med. Rafala Masztaka, Warsaw
  - EMC Instytut Medyczny SA, Wroclaw
- Portugal (7):
  - ULSM - Hospital Pedro Hispano, Matosinhos Municipality, Porto District
  - Unidade Local de Saude Almada-Seixal | Hospital Garcia de Orta - Research Department, Almada, Setúbal District
  - IPO Lisboa, Lisbon
  - CHLC - Hospital Sao Jose, Lisbon
  - Luz Saude | Hospital da Luz Lisboa - Centro de Investigacao Clinica, Lisbon
  - IPO Porto, Porto
  - Centro Hospitalar Universitario de Sao Joao | Polo Porto - Centro de Investigacao e Ensaios Clinicos, Porto
- Romania (4):
  - Institutul Clinic Fundeni, Bucharest
  - Sf. Nectarie Oncology Center, Craiova
  - Spitalul Clinic Judetean de Urgenta Oradea, Oradea
  - Spitalul Clinic Judetean Mures, Târgu Mureş
- Russia (20):
  - Ltd "EVIMED", Chelyabinsk
  - Chelyabinsk Regional Oncology Dispensary, Chelyabinsk
  - Ivanovo Regional Oncology Dispensary, Ivanovo
  - Republican Clinical Oncology Dispensary Kazan, Kazan'
  - Krasnoyarsk Regional Clinical Oncology Dispensary, Krasnoyarsk
  - Russian Oncological Scientific Center n.a. N.N. Blokhin RAMS, Moscow
  - Moscow Scient. Res. Institute of Oncology n.a P.A. Hertzen, Moscow
  - City clinical hospital #40 Moscow, Moscow
  - City Outpatient Clinic #1 of Privolzhsky Regional Med. Cent., Nizhny Novgorod
  - LLC Reafan, Novosibirsk
  - Medical Center "Avicenna", Novosibirsk
  - National Medical Research Radiology Center, Obninsk
  - Clinical Oncological Dispensary of Omsk Region, Omsk
  - Rostov State Medical University, Rostov-on-Don
  - Leningrad Regional Oncology Dispensary, Saint Petersburg
  - St. Petersburg Clinical Hospital of RAS, Saint Petersburg
  - St. Petersburg Medical University n.a. I.P. Pavlov, Saint Petersburg
  - Saratov State Medical University, Saratov
  - Multi-Field Clinical Medical Center "Medical City", Tyumen
  - Regional Clinical Oncology Dispensary, Vladimir
- Serbia (2):
  - Clinical Hospital Center Bezanijska kosa, Belgrade
  - Clinical Center Nis, Niš
- Slovakia (3):
  - J. BREZA MEDICAL s. r. o., Bratislava
  - CUIMED s.r.o, Bratislava
  - Privatna urologicka ambulancia, s.r.o., Trenčín
- South Africa (6):
  - Cancercare Outeniqua, George, Eastern Cape
  - Langehoven Drive Oncology Centre, Port Elizabeth, Eastern Cape
  - University of Pretoria, Clinical Research Unit, Pretoria, Gauteng
  - Dept Radiation and Oncology Tygerberg Academic Hospital, Cape Town, Western Cape
  - Cape Gate Oncology Centre, Cape Town, Western Cape
  - Cancercare Rondebosch Oncology, Rondebosch, Western Cape
- South Korea (13):
  - Chonnam National University Hospital, Gwangju, Gwangju Gwang''yeogsi
  - Seoul National Univ. Bundang Hospital, Seongnam-si, Gyeonggido
  - Chungbuk National University Hospital, Cheongju-si, North Chungcheong
  - Severance Hospital, Yonsei University Health System, Seoul, Seoul Teugbyeolsi
  - Asan Medical Center - Oncology Department, Seoul, Seoul Teugbyeolsi
  - Seoul National University Hospital, Seoul, Seoul Teugbyeolsi
  - Gangnam Severance Hospital, Yonsei University Health System, Seoul, Seoul Teugbyeolsi
  - Inje University Busan Paik Hospital, Busan
  - Keimyung University Dongsan Medical Center, Daegu
  - Kyungpook National University Chilgok Hospital, Daegu
  - Gachon University Gil Medical Center, Incheon
  - Samsung Medical Center - Oncology Department, Seoul
  - The Catholic University of Korea Seoul St. Mary's Hospital, Seoul
- Spain (24):
  - Hospital General de Elche - Urologia, Elche, Alicante
  - Parc Tauli Hospital Universitari - Oncologia, Sabadell, Barcelona
  - Hospital SAS de Jerez de la Frontera, Jerez de la Frontera, Cádiz
  - Hospital de Manacor - Urologia, Manacor, Illes Baleares
  - Hospital Universitari Son Espases - Oncologia, Palma de Mallorca, Illes Baleares
  - Hospital Universitario Fundacion Alcorcon - Urologia, Alcorcón, Madrid
  - Hospital del Mar, Barcelona
  - Ciutat Sanitaria i Universitaria de la Vall d'Hebron, Barcelona
  - Hospital Clínic i Provincial de Barcelona, Barcelona
  - Hospital de la Santa Creu i de Sant Pau | Oncología, Barcelona
  - Hospital Universitari de Bellvitge (HUB), Barcelona
  - Hospital San Pedro de Alcántara - Oncologia, Cáceres
  - Hospital Universitario Reina Sofia - Oncologia, Córdoba
  - Hospital Universitario Lucus Augusti - Urologia, Lugo
  - Hospital General Universitario Gregorio Maranon | Oncologia, Madrid
  - Hospital Universitario Ramon Y Cajal - Oncologia, Madrid
  - Hospital Clinico Universitario San Carlos | Oncologia, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Virgen De La Victoria - Oncology, Málaga
  - Hospital Clínico de Salamanca, Salamanca
  - Hospital Universitario Virgen Del Rocio S.L. - Oncologia, Seville
  - Instituto Valenciano de Oncología, Valencia
  - Hospital Arnau De Vilanova De Valencia - Oncologia, Valencia
- Sweden (5):
  - Sahlgrenska Universitetssjukhuset, Gothenburg
  - Skånes Universitetssjukhus Malmö, Malmo
  - Karolinska Universitetssjukhuset, Stockholm
  - Norrlands Universitetssjukhus, Umea, Umeå
  - Akademiska Sjukhuset, Uppsala
- Taiwan (6):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Kaohsiung
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital at Linkou, Taoyuan District
- Turkey (Türkiye) (2):
  - Gazi Universitesi Tip Fakultesi, Ankara
  - TC Saglik Bakanligi Goztepe ProfDr Suleyman Yalcin Sehir Has, Istanbul
- Ukraine (7):
  - CNE "Clinical Center of Oncology, Hematology, Transplantology and Palliative Care of the Cherkasy Regional Council", Cherkasy
  - Regional communal non-profit enterprise 'Chernivtsi regional clinical hospital' - Urological department, Chernivtsi
  - Municipal Non-commercial Enterprise 'City Clinical Hospital #4' of Dnipro City Council - City ?hemotherapy ?enter, Dnipro
  - Regional Medical Clinical Center of Urology and Nephrology n.a. V. I. Shapoval - Department of Oncologic Urology #5, Kharkiv
  - Kyiv City Hospital #3 - Department of Urology, Kyiv
  - SE "Academician O.F. Vozianov Institute of Urology" of NAMSU - Division of Reconstructive Urology and Advanced Technologies, Kyiv
  - Zakarpattia Anti-Tumor Centre - Chemotherapy Department, Uzhhorod
- United Kingdom (12):
  - Royal Berkshire NHS Foundation Trust¦Royal Berkshire Hospital - Oncology, Reading, Berkshire
  - Prince Philip Hospital, Llanelli, Carmarthenshire
  - East Suffolk and North Essex NHS Foundation Trust¦Colchester General Hospital - Oncology Trials Unit, Colchester, Essex
  - Clatterbridge Centre for Oncology, Bebington, Merseyside
  - Scunthorpe General Hospital, Scunthorpe, North East Lincolnshire
  - Dudley Group NHS Foundation Trust ¦Russells Hall Hopsital - Oncology, Dudley, West Midlands
  - Calderdale and Huddersfield NHS Foundation Trust¦Huddersfield Royal Infirmary - Oncology, Huddersfield, West Yorkshire
  - Mid Yorkshire Teaching NHS Trust¦Pinderfields Hospital - Oncology, Wakefield, West Yorkshire
  - Cardiff and Vale University Health Board | University Hospital of Wales - Nephrology and Transplant, Cardiff
  - NHS Greater Glasgow & Clyde | Beatson West of Scotland Cancer Centre - Clinical Research Unit, Glasgow
  - University College London Hospitals NHS Foundation Trust, London
  - Charing Cross Hospital, London

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.